CLINICAL TRIAL: NCT05640284
Title: Evaluation of the Effect of Periimplant Soft Tissue Phenotype on Marginal Bone Loss Using Biochemical Approach
Brief Title: Evaluation of the Effect of Periimplant Soft Tissue Phenotype on Marginal Bone Loss
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Zeynep Tastan Eroglu, assistant professor, Necmettin Erbakan University
Other Study IDs: periimplantmicrorna
Record Dates: First submitted 2022-11-25; First posted 2022-12-07 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Alveolar Bone Loss; Dental Implant; Periimplantitis
Keywords: periimplantitis; MicroRNA; dental implants; soft tissue phenotype; alveolar bone loss
MeSH Terms: conditions — Alveolar Bone Loss; Peri-Implantitis | interventions — Radiography, Panoramic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Adequate KMT: Keratinized mucosal thicknesses (KMT) on their buccal surfaces are 2 mm and above.
  Interventions: Diagnostic Test: Nuclear Factor-Kappa B Ligand (RANKL) analysis; Diagnostic Test: Osteoprotegerin (OPG) analysis; Diagnostic Test: Tumor Necrosis Factor Alpha (TNF-α) analysis; Diagnostic Test: MicroRNA-223 analysis; Diagnostic Test: Microrna-27a analysis
- inadequate KMT: Keratinized mucosal thicknesses (KMT) on their buccal surfaces are less than 2 mm.
  Interventions: Diagnostic Test: Nuclear Factor-Kappa B Ligand (RANKL) analysis; Diagnostic Test: Osteoprotegerin (OPG) analysis; Diagnostic Test: Tumor Necrosis Factor Alpha (TNF-α) analysis; Diagnostic Test: MicroRNA-223 analysis; Diagnostic Test: Microrna-27a analysis
- adequate KGW: keratinized gingival width (KGW) on their buccal surfaces are 2 mm and above.
  Interventions: Diagnostic Test: Nuclear Factor-Kappa B Ligand (RANKL) analysis; Diagnostic Test: Osteoprotegerin (OPG) analysis; Diagnostic Test: Tumor Necrosis Factor Alpha (TNF-α) analysis; Diagnostic Test: MicroRNA-223 analysis; Diagnostic Test: Microrna-27a analysis
- inadequate KGW: keratinized gingival width (KGW) on their buccal surfaces are less than 2 mm.
  Interventions: Diagnostic Test: Nuclear Factor-Kappa B Ligand (RANKL) analysis; Diagnostic Test: Osteoprotegerin (OPG) analysis; Diagnostic Test: Tumor Necrosis Factor Alpha (TNF-α) analysis; Diagnostic Test: MicroRNA-223 analysis; Diagnostic Test: Microrna-27a analysis
- Peri-implant health: The absence of signs of inflammation (redness, swelling, bleeding on probing) in the peri-implant soft tissue, probing depth (PD) ≤5 mm with mild force (approximately 0.25 N), and no further bone loss following initial healing are defined as "peri-implant health".
  Interventions: Diagnostic Test: Nuclear Factor-Kappa B Ligand (RANKL) analysis; Diagnostic Test: Osteoprotegerin (OPG) analysis; Diagnostic Test: Tumor Necrosis Factor Alpha (TNF-α) analysis; Diagnostic Test: MicroRNA-223 analysis; Diagnostic Test: Microrna-27a analysis
- peri-implant mucositis: "Peri-implant mucositis" is defined as clinically observable signs of inflammation (swelling, redness and soft consistency of tissue), bleeding on probing (lines or drops) and/or signs of suppuration in the absence of bone loss greater than 2 mm, the threshold for initial bone remodulation.
  Interventions: Diagnostic Test: Nuclear Factor-Kappa B Ligand (RANKL) analysis; Diagnostic Test: Osteoprotegerin (OPG) analysis; Diagnostic Test: Tumor Necrosis Factor Alpha (TNF-α) analysis; Diagnostic Test: MicroRNA-223 analysis; Diagnostic Test: Microrna-27a analysis

INTERVENTIONS:
Diagnostic Test: Nuclear Factor-Kappa B Ligand (RANKL) analysis — samples of peri-implant groove fluid will be taken with paper strips and RANKL assessment will be made
Diagnostic Test: Osteoprotegerin (OPG) analysis — samples of peri-implant groove fluid will be taken with paper strips and OPG assessment will be made
Diagnostic Test: Tumor Necrosis Factor Alpha (TNF-α) analysis — samples of peri-implant groove fluid will be taken with paper strips and TNF-α assessment will be made
Diagnostic Test: MicroRNA-223 analysis — samples of peri-implant groove fluid will be taken with paper strips and MicroRNA-223 assessment will be made
Diagnostic Test: Microrna-27a analysis — samples of peri-implant groove fluid will be taken with paper strips and Microrna-27a assessment will be made

SUMMARY:
The goal of this clinical trial to test the effect of periimplant soft tissue phenotype in the participants with implant placed and at least 1 year after implant loading. The main questions it aims to answer are:

1. Is keratinized mucosal thickness (KMT) important in early marginal bone loss and peri implant health?
2. Is keratinized gingival width (KGW) important in early marginal bone loss and and peri implant health? The researchers plan to include 80 implants in the study. These 80 implants will be divided into 2 groups in 2 different ways according to their KMT and KGW on their buccal surfaces: KMT ≥2 mm are included in the adequate KMT, and those with KMT<2 mm are in the insufficient KMT group. Those with KGW≥2 mm are adequate KGW, those with KGW<2 mm are adequate KGW. The researchers will assess marginal bone loss around the implant using radiographs and collect peri-implant crevicular fluid (PICF) using paper strips. Another researchers will measure the Receptor Activator Of Nuclear Factor-Kappa B Ligand (RANKL), Osteoprotegerin (OPG), Tumor Necrosis Factor Alpha (TNF-α), MicroRNA-223 (MiRNA-223), MicroRNA-27a (MiRNA-27a) levels in the collected PICF. They will compare radiographic bone loss and biomarker levels in groups.

DETAILED DESCRIPTION:
Early marginal bone loss around the implant can be caused by various reasons. Keratinized mucosal thickness (KMT) and keratinized gingival width (KGW) are components of periimplant soft tissue. Recently, KGW and KMT in the peri-implant region have been investigated as possible factors influencing this phenomenon.

The hypothesis of this study: Periimplant soft tissue phenotype is associated with marginal bone loss and peri implant health through Receptor Activator Of Nuclear Factor-Kappa B Ligand (RANKL), Osteoprotegerin (OPG), Tumor Necrosis Factor Alpha (TNF-α), MicroRNA-223 (MiRNA-223) and Microrna-27a 80 implants, at least 1 year after their loading, in patients who continued their routine controls will be included in the study. The participants in this study were selected from patients who underwent implant placement by the same periodontologist (E.Ö.) in the Department of Periodontology of Necmettin Erbakan University in 2020 and still have 6-month radiographic and clinical follow-up. Selected patients, those who signed the written informed consent form were included in the study. In the study, the first radiographs of all patients, the clinical and radiographic conditions obtained at the 6-month routine control examination will be evaluated. During the same routine controls, a sample of peri-implant groove fluid was taken with paper strips.

Diagnoses of the implants included in the study will be made using the criteria of the 2017 World Workshop on Periodontal and Peri-implant Diseases and Conditions. 2 mm marginal bone loss (MBL) which may occur during the bone remodeling process after implant placement and loading, is accepted as the threshold. The absence of signs of inflammation (redness, swelling, bleeding on probing) in the peri-implant soft tissue, probing depth (PD) ≤5 mm with mild force (approximately 0.25 N), and no further bone loss following initial healing are defined as "periimplant health". "Peri-implant mucositis" is defined as clinically observable signs of inflammation (swelling, redness and soft consistency of tissue), bleeding on probing (BOP) (lines or drops) and/or signs of suppuration in the absence of bone loss greater than 2 mm, the threshold for initial bone remodulation defined. The definition of "peri-implantitis" is clinically observable signs of inflammation, probing bleeding and/or suppuration, increased probing depth, progressive bone loss after implant restoration, or MBL ≥3 mm with profuse bleeding in the absence of initial radiographs and PD was ≥6 mm. Implants with periimplantitis will be excluded. Implants will be divided into 2 groups according to their peri-implant health: Peri-implant health and peri-implant mucositis.

In addition to routine clinical and radiographic examination of the implants, KMT and KGW measurements will be made. they will be divided into 2 groups in 2 ways. According to KMT on their buccal surfaces: KMT ≥2 mm are included in the adequate KMT, and those with KMT <2 mm are in the inadequate KMT group (60). According to KGW on their buccal surfaces: KGW≥2 mm are adequate KGW, those with KGW<2 mm are inadequate KGW.

Radiographic evaluation will be made using intraoral periapical radiographs obtained using the parallel technique with the plastic film holder. Calibration of digital images will be performed using the length of the implant as a well-defined fixed reference point. The bone level measurement will be made by measuring between the bone-implant first contact point and the reference point in the coronal part of the implant body selected for different implant systems in both the mesial and distal directions of the implants. In order to evaluate the marginal bone loss (MBL), the measurements obtained will be compared with the measurements on the radiographs taken after the delivery of the prosthesis.

Peri-implant crevicular fluid (PIGF) will be collected from the participants for the biochemical evaluation to be made. PIGF specimens will be collected from the mesiobuccal of each implant, prior to any periodontal probing, and after removal of the supra mucosal plate. The area to be sampled will be insulated with cotton rolls and air-dried. The paper will be advanced with the strip until it shows slight resistance and held in the sample area for 30 seconds. Samples will be stored at -70˚C.

TNF-α, RANKL, OPG and MiRNA 223 and MiRNA 27a evaluations of the peri-implant crevicular fluid (PIGF) collected from the patients will be performed. TNF-α, RANKL and OPG will be evaluated by the Enzyme-Linked ImmunoSorbent Assay (ELISA) method. MiRNA 223 and MiRNA 27a evaluations will be performed using Real-Time Polymerase Chain Reaction (RT-PCR).

Marginal bone loss and biomarker levels will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one fixed restoration on a titanium dental implant in the mouth
* Over-implant restoration, functioning for at least 12 months
* Attending our preventive care regularly (≥1/year)
* Non-smokers

Exclusion Criteria:

* Receiving head or neck radiation in the last 6 months
* Bisphosphonate users
* Those who have received antibiotic treatment in the last 3 months
* Patients with diabetes mellitus (hemoglobin A1c ≥7.0) that may affect the outcome of implant therapy
* implants with peri-implantitis
* Pregnant or breastfeeding mothers
* Those with metabolic bone disorders
* Those who have a history of periodontitis and have undergone any periodontal treatment in the last year
* Those whose implant positions are not suitable
* Implants using soft or hard tissue grafts before, during, or after implant placement
* Those with a restoration that did not allow accurate probing depth recording were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participants will be selected from among the patients whose implant placement was performed by the same periodontologist (E.Ö) at Necmettin Erbakan University, Department of Periodontology between 2020 and whose radiographic and clinical follow-up is still ongoing for 6 months. Of each selected study patient, those who signed the written informed consent form and met the inclusion and exclusion criteria will be included in the study.
  80 implants in approximately 40 patients are planned to be included in the trial.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Comparison of mean Receptor Activator Of Nuclear Factor-Kappa B Ligand (RANKL) level between peri-implant health and peri-implant mucositis groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The RANKL levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via Enzyme-Linked ImmunoSorbent Assay . The difference between the groups will be evaluated.
Comparison of mean Osteoprotegerin (OPG) level between peri-implant health and peri-implant mucositis groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The OPG levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via Enzyme-Linked ImmunoSorbent Assay . The difference between the groups will be evaluated.
Comparison of mean Tumor Necrosis Factor Alpha (TNF-α) level between peri-implant health and peri-implant mucositis groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The TNF-α levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via Enzyme-Linked ImmunoSorbent Assay . The difference between the groups will be evaluated.
Comparison of mean MicroRNA-223 level between peri-implant health and peri-implant mucositis groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The MicroRNA-223 levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via real-time polymerase chain reaction. The difference between the groups will be evaluated.
Comparison of mean MicroRNA-27a level between peri-implant health and peri-implant mucositis groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The MicroRNA-27a levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via real-time polymerase chain reaction. The difference between the groups will be evaluated.
Comparison of alveolar bone loss between adequate Keratinized mucosal thickness (KMT) and inadequate KMT groups | It will be done at the start of the study, immediately after the control radiograph is taken.
  The bone level measurement will be made by measuring between the bone-implant first contact point and the reference point in the coronal part of the implant body selected for different implant systems in both the mesial and distal directions of the implants. In order to evaluate the marginal bone loss (MBL), the measurements obtained will be compared with the measurements on the radiographs taken after the delivery of the prosthesis.
Comparison of alveolar bone loss between between adequate keratinized gingival width (KGW) and inadequate KGW groups | It will be done at the start of the study, immediately after the control radiograph is taken.
  The bone level measurement will be made by measuring between the bone-implant first contact point and the reference point in the coronal part of the implant body selected for different implant systems in both the mesial and distal directions of the implants. In order to evaluate the marginal bone loss (MBL), the measurements obtained will be compared with the measurements on the radiographs taken after the delivery of the prosthesis.
Comparison of mean Receptor Activator Of Nuclear Factor-Kappa B Ligand (RANKL) level between adequate KMT and inadequate KMT groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The RANKL levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via Enzyme-Linked ImmunoSorbent Assay . The difference between the groups will be evaluated.
Comparison of mean Receptor Activator Of Nuclear Factor-Kappa B Ligand (RANKL) level between adequate KGW and inadequate KGW groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The RANKL levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via Enzyme-Linked ImmunoSorbent Assay . The difference between the groups will be evaluated.
Comparison of mean Osteoprotegerin (OPG) level between adequate Keratinized mucosal thickness (KMT) and inadequate KMT groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The OPG levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via Enzyme-Linked ImmunoSorbent Assay . The difference between the groups will be evaluated.
Comparison of mean Osteoprotegerin (OPG) level between between adequate keratinized gingival width (KGW) and inadequate KGW groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The OPG levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via Enzyme-Linked ImmunoSorbent Assay . The difference between the groups will be evaluated.
Comparison of mean Tumor Necrosis Factor Alpha (TNF-α) level between adequate Keratinized mucosal thickness (KMT) and inadequate KMT groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The TNF-α levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via Enzyme-Linked ImmunoSorbent Assay . The difference between the groups will be evaluated.
Comparison of mean Tumor Necrosis Factor Alpha (TNF-α) level between between adequate keratinized gingival width (KGW) and inadequate KGW groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The TNF-α levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via Enzyme-Linked ImmunoSorbent Assay . The difference between the groups will be evaluated.
Comparison of mean MicroRNA-223 level between adequate Keratinized mucosal thickness (KMT) and inadequate KMT groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The MicroRNA-223 levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via real-time polymerase chain reaction. The difference between the groups will be evaluated.
Comparison of mean MicroRNA-223 level between between adequate keratinized gingival width (KGW) and inadequate KGW groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The MicroRNA-223 levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via real-time polymerase chain reaction. The difference between the groups will be evaluated.
Comparison of mean MicroRNA-27a level between adequate Keratinized mucosal thickness (KMT) and inadequate KMT groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The MicroRNA-27a levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via real-time polymerase chain reaction. The difference between the groups will be evaluated.
Comparison of mean MicroRNA-27a level between between adequate keratinized gingival width (KGW) and inadequate KGW groups | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The MicroRNA-27a levels in the peri-implant crevicular fluid (PIGF) collected from the patients will be measured via real-time polymerase chain reaction. The difference between the groups will be evaluated.

SECONDARY OUTCOMES:
Correlation between MBL amounts and TNF-α | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The correlation MBL amounts and TNF-α will be evaluated.
Correlation between MBL amounts and RANKL | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The correlation MBL amounts and RANKL will be evaluated.
Correlation between MBL amounts and OPG | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The correlation MBL amounts and OPG will be evaluated.
Correlation between MBL amounts and MicroRNA-223 | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The correlation MBL amounts and MicroRNA-223 will be evaluated.
Correlation between MBL amounts and MicroRNA-27a | this will be done at the beginning of the study, after samples have been collected from all implants in the study.
  The correlation MBL amounts and MicroRNA-27a will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: zeynep taştan eroğlu, Study Director — Necmettin Erbakan University; dilek özkan şen, Principal Investigator — Necmettin Erbakan University; elif öncü, Principal Investigator — Lokman Hekim University
Locations (1):
- Necmettin Erbakan University, dentistry Faculty, Konya, Turkey (Türkiye)